CLINICAL TRIAL: NCT00440232
Title: A Pilot Trial Examining the Safety and Efficacy of Frovatriptan as a Preemptive Treatment for Fasting-Induced Migraine Headache
Brief Title: A Research Study To Evaluate If Frovatriptan Is Safe And Effective In Preventing Migraine Headache After Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Stephen D. Silberstein, M.D., Jefferson Headache Center, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDS/FHA-FRV/ 01
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — frovatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Frovatriptan (Experimental): 5.0 mg of Frovatriptan given as single dose
  Interventions: Drug: Frovatriptan
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Frovatriptan — Frovatriptan 5.0 mg orally one time at the start of the 20 hour fast
  Other Names: Frova
  Arms: Frovatriptan
Drug: Placebo — Inert tab identical in appearance to Frovatriptan
  Arms: placebo

SUMMARY:
We are testing the hypothesis that subjects in the treatment group will experience fewer fasting induced headaches as compared to those in the placebo group.In our clinical experience, we estimate that approximately 25% of our headache population experiences fasting-induced migraine or hunger-induced migraine. With a given migraine incidence of 28 million in the United States alone, we estimate that approximately 7 million will experience hunger as a migraine trigger. If an individual has a known migraine trigger, then there are a variety of ways to modify care in order to address that trigger. The simplest is to avoid that trigger or preemptively treat that trigger. Frovatriptan has good evidence for daily use for a short time to help prevent menstrually related migraines. A short course of treatment can often avoid the initiation of the migraine and improve quality of life. Knowing that a longer acting triptan, such as frovatriptan, has demonstrated capability at suppressing headache through a known trigger, suggests the need to study this with fasting induced migraines, as well.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65, inclusive
* Subjects diagnosed with episodic migraine, with or without aura according to IHS criteria for at least one-year prior to screening
* Subjects who experience between 1 and 6 migraine attacks per month inclusive (during the previous 6 months) with no more than 15 days of headache per month.
* Subject reports hunger or fasting as a known trigger for migraine
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Subjects who are able to understand and comply with all study procedures.
* Subject is willing to complete one 20-hour fast, starting between 5:00 and 8:00 P.M., with no food or drink (except water needed to take routine medication)
* Subject provides written informed consent prior to any screening procedures being conducted
* If subject is taking a preventive migraine medication for migraine or any other reason, that medication must have been a stable dose for at least 4 weeks prior to screening, and must remain stable throughout the duration of the study.

EXCLUSION CRITERIA

* Pregnant and/or lactating women
* Subjects who have a history of clinically relevant allergy to frovatriptan or like compounds
* Subjects who, in the investigators opinion, have a history or have evidence of any other medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects who currently have or have a history of significant cerebrovascular disease including basilar or hemiplegic migraine
* Subjects who have a history of non-response to triptans, as determined by investigator
* Subjects with uncontrolled hypertension
* Subjects with diabetes mellitus who require insulin or oral anti-hyperglycemic agents will be excluded. (Subjects with Type II diabetes who are well controlled with diet and exercise alone may be included.)
* Subjects who currently have or who have a history of ischemia and/or vasospastic coronary artery disease
* Subjects who, in the investigators opinion, have significant risk factors of coronary artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Silberstein, M.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from our office practice or surrounding community from 7/16/07 through 3/18/09
Period: Overall Study
Arm/Group | Frovatriptan | Placebo
Started | 36 | 38
Completed | 33 | 34
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Unable to treat within allowed time | 0 | 1
Not completed — Onset of headache within 4 hours of fast | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Frovatriptan | Placebo | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 38 | 74
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.15 (11.8) | 38.7 (12.7) | 39.49 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Fasting-induced Headache of Any Intensity
Description: Incidence of fasting-induced headache of any intensity occurring at greater than 4 hours, but within 20 hours after onset of fasting
Time Frame: 20 hours
Measure: Number; unit: participants
Arm/Group | Frovatriptan | Placebo
Number analyzed (Participants) | 33 | 34
participants | 12 | 18
Statistical Analysis 1: Comparison: Frovatriptan vs Placebo; Test type: Superiority or Other; p = 0.172, Chi-squared; Odds Ratio (OR) = 1.969, 95% CI 2-sided [0.74 to 5.235]

2. Secondary Outcome: Time to Development of Headache of Any Intensity
Description: Time to development of headache of any intensity in the 2 treatment arms
Time Frame: 20 hours
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Frovatriptan | Placebo
Number analyzed (Participants) | 33 | 34
hours | 17.388 [16.05 to 18.73] | 17.06 [15.72 to 18.40]
Statistical Analysis 1: Comparison: Frovatriptan vs Placebo; Test type: Superiority or Other; p = 0.264, Log Rank; df=1; log rank chi square = 1.247

ADVERSE EVENTS:
Arm/Group | Frovatriptan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 1/35 | 5/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Frovatriptan (N=35) | Placebo (N=36)
nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) — Nausea (may be secondary to study medication or associated symptom of migraine)
sleepiness/fatigue (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes